CLINICAL TRIAL: NCT02104050
Title: A Phase 2b Randomized, Double-Blind, Vehicle-Controlled, Repeat-Dose, Multi- Center, Efficacy and Safety Clinical Trial of Topically Applied OLT1177 Gel in Subjects With Moderate to Severe Pain Associated With Osteoarthritis of the Knee Following Cessation of Pain Therapy
Brief Title: Study of OLT1177 Gel to Treat Moderate to Severe OA Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OLT1177-03
Record Dates: First submitted 2014-03-28; First posted 2014-04-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo Gel (Placebo Comparator): 6 mL of Placebo Gel administered TID for 6 weeks
  Interventions: Drug: Placebo Gel
- OLT1177 Gel (Experimental): 6 mL of OLT1177 Gel (5%) administered TID for 6 weeks
  Interventions: Drug: OLT1177 Gel

INTERVENTIONS:
Drug: Placebo Gel — 6 mL of Placebo Gel administered TID for 6 weeks
  Arms: Placebo Gel
Drug: OLT1177 Gel — 6 mL of OLT1177 Gel (5%) administered TID for 6 weeks
  Arms: OLT1177 Gel

SUMMARY:
The objectives of this trial are to investigate the efficacy and safety of six weeks of treatment with OLT1177 Gel in subjects with moderate to severe pain associated with osteoarthritis of the knee following cessation of pain therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 80 years old, inclusive
* Clinical diagnosis of osteoarthritis in one target knee based on the following American College of Rheumatology (ACR) criteria:

  1. Knee Pain
  2. At least 1 of 3:

     * Age > 50 years
     * Morning stiffness lasting < 30 minutes
     * Crepitus on motion
  3. Osteophytes on radiograph
* Symptoms associated with osteoarthritis of the knee (including pain) for ≥ 6 months prior to Screening
* Knee pain associated with osteoarthritis, which required NSAID or other therapy for ≥ 15 days during the preceding month
* Radiographic evidence of osteoarthritis by Kellgren-Lawrence classification with a rating of Grade 2 or 3 in the target knee (does not include borderline Grade 2), as confirmed by the Sponsor's designated rheumatologist through radiographic review of x-ray(s) taken no more than 1 year prior to the Screening visit. (Sharpening of the tibial spine is not considered to be an osteophyte) (See Appendix 4 for additional details)
* Meets pain assessment entry criteria as defined by Sponsor's pain eligibility algorithm and calculated by the study Interactive Web Response System
* No clinically significant change in physical activity and/or therapy for the past 3 months
* Able to provide written informed consent prior to initiation of any clinical trial-related procedures; and willing and able, in the opinion of the Investigator, to comply with all requirements of the clinical trial for the duration of the trial (such requirements include, but are not limited to: attending all study visits, refraining from elective surgery or extensive travel during participation)

Exclusion Criteria:

General

* Women of childbearing potential, or men whose sexual partner(s) is a woman of childbearing potential may not be entered into the study if:

  1. They are or intend to become pregnant (including use of fertility drugs) during the study
  2. They are nursing
  3. They are not using an acceptable, highly effective method of contraception until all follow-up procedures are complete. (Acceptable, highly effective forms of contraception are defined as: oral contraception, intrauterine device, systemic [injectable or patch] contraception, double barrier methods, naturally or surgically sterile, strict abstinence or partner has been sterilized. If hormonal-based birth control is being used, subject or subject's sexual partner(s) must be on a stable-dose for ≥ 3 months prior to the Baseline visit and maintained at the same dosing level throughout the 9-week clinical trial.)
* Body Mass Index (BMI) over 40
* A history of osteoarthritis symptoms that are completely non-responsive to non-steroidal anti-inflammatory drugs (NSAIDs) at the discretion of the Investigator
* Planned change (increase or decrease) in subject's level of physical activity (e.g., aerobic or anaerobic exercise) during the 6-week Treatment Period following randomization
* Enrollment in any trial and/or use of any Investigational Drug or device within the immediate 30-day period prior to the Baseline visit
* Enrollment in any study previously sponsored by Olatec Industries LLC, specifically Study OLT1177-01 or OLT1177-02

Pain Related

* Does not meet pain assessment entry criteria as defined by Sponsor's pain eligibility algorithm and calculated by the study Interactive Web Response System
* Clinically significant joint (other than the knee) or general pain at Baseline, at the discretion of the Investigator

Musculoskeletal Related

* Clinically significant, excessive effusion heat and/or redness in the target knee as determined by the Investigator
* Knock-kneed or bow-legged, as defined by a valgus or varus deformity of ≥ 15 degrees
* Radiographic evidence of osteoarthritis by Kellgren-Lawrence classification with a rating of Grade 0, 1 or 4 in the target knee, as confirmed by the Sponsor's designated rheumatologist through radiographic review of x-ray(s) taken no more than 1 year prior to the Screening visit (sharpening of the tibial spine is not considered to be an osteophyte)
* Documented history of clinically significant pain associated with osteoarthritis of the spine or hips, at the discretion of the Investigator
* Significant anterior knee pain due to diagnosed isolated patella-femoral syndrome or chondromalacia
* Clinically significant medio-lateral and/or anterior-posterior instability, at the discretion of the Investigator
* Open surgery of the target knee within the prior year or surgery to the contralateral knee or other weight-bearing joint within the prior year, if at the discretion of the Investigator it would interfere with the study. If subject had open surgery more than one-year prior, Sponsor's designated rheumatologist must confirm that such surgery did not have any negative impact or consequence to the target knee (e.g., deformity of angle to the bone, bone on bone, locking joints, etc.)
* Arthroscopic surgery of the target knee within the prior six months
* Any acute or chronic injury, other than osteoarthritis in the target knee, that will be treated during the trial with any medication not allowed during the Treatment Period
* Prior surgery of the target knee requiring insertion of a medical device or surgical hardware (e.g., screws)
* Any major trauma or injury (including sports injuries) to the target knee in the past 12 months
* Documented history of inflammatory joint disease, including but not limited to: rheumatoid arthritis, gout, pseudogout, Paget's disease, psoriatic arthritis, ankylosing spondylitis, chronic inflammatory disease (e.g., colitis), fibromyalgia (diagnosed in accordance with ACR criteria, as applicable), articular fracture, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary osteochondromatosis, heritable disorders (e.g., hypermobility) or collagen gene mutations
* Any planned interventional and/or surgical procedure during the 6-week Treatment Period following randomization

Concomitant Conditions, Diseases, Medications/Therapies and Medical History Related

* Any use of Rescue Medication within 24 hours prior to the Baseline visit or use of any other pain medication within 7 days prior to Baseline visit
* Uncontrolled hypertension, defined as blood pressure ≥ 150/95 mmHg
* A history of uncontrolled and untreated diabetes mellitus with an HbA1c level > 8; or blood sugar levels that are outside of the normal range and HbA1c level > 8 is subsequently confirmed
* Any inflammatory skin condition over the target knee application area
* Use of any prohibited concomitant medications/therapies during the 7-day Washout Period or planned use of any prohibited concomitant medications/therapies during the 6 week Treatment Period
* Use of intraarticular or intramuscular steroids in the target knee within the previous 3 months or in any other joint within the previous 30 days
* Use of intraarticular hyaluronate in the target knee within the previous 6 months or in any other joint within the previous 30 days
* Current substance abuse or history of chronic substance abuse within the past year, or prior chronic substance abuse (including alcoholism and/or addiction to pain medications) that is determined at the discretion of the Investigator as likely to interfere with trial assessments or recur during the trial
* Use of any systemic (oral or parenteral) corticosteroids within the prior month
* Uncontrolled psychiatric conditions (e.g., mania, depression, anxiety, substance dependence of any kind) that would impair the subject from safely participating in the trial, including completing any protocol requirements
* Evidence of cognitive impairment including dementia that may interfere with subject's ability to complete daily pain diaries requiring recall of average pain level in the past 24 hours
* Significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological or neurological disease or prior surgery that may interfere with the subject successfully completing the trial, including completing any protocol requirements as determined by the Investigator
* History of or known positive for HIV, Hepatitis B surface antigen (HBsAg) or antibodies to Hepatitis C Virus (HCV)
* Diagnosed with any form of cancer within the past 5 years, except for treated basal cell or squamous cell carcinoma of the skin
* Any other medical conditions, diseases or prior surgeries that in the opinion of the Investigator would impair the subject from safely participating in the trial and/or completing any protocol requirements
* Active infection within 3 days of the Baseline visit

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain on Movement | Baseline to Week 6
  Subjects will record their level of Pain on Movement in the target knee on a 100-mm VAS scale (with anchors 0=no pain; 100=extreme pain) in response to the question, 'How do you estimate the average amount of your study knee pain while moving during your daily activities within the last 24 hours?'

SECONDARY OUTCOMES:
Current Knee Pain | Baseline (pre-dose) to Baseline (50-min post-dose)
  After completing a walk of approximately 50 feet, subjects will record their level of Current Knee Pain in the target knee on a 100-mm Visual Analog Scale (with anchors 0=no pain; 100=extreme pain) in response to the question, 'How do you estimate the amount of your study knee pain right now?'
WOMAC Pain Subscale | Baseline to Weeks 2, 4 and 6
  The WOMAC NRS3.1 OA Index is a validated, segregated, multidimensional, self-administered index with three independent dimensions: pain, physical function and stiffness. It is comprised of 24 questions to be answered by the subject. The pain subscale consists of 5 questions; the physical function subscale consists of 17 questions; and the joint stiffness subscale consists of 2 questions.
WOMAC Physical Function Subscale | Baseline to Weeks 2, 4 and 6
  The WOMAC NRS3.1 OA Index is a validated, segregated, multidimensional, self-administered index with three independent dimensions: pain, physical function and stiffness. It is comprised of 24 questions to be answered by the subject. The pain subscale consists of 5 questions; the physical function subscale consists of 17 questions; and the joint stiffness subscale consists of 2 questions.
Global Rating of Disease | Baseline to Weeks 2, 4 and 6
  Subjects will complete the assessment on a 100-mm Visual Analog Scale (with anchors 0=very good; 100=very poor) in response to the question, 'Considering all the ways osteoarthritis affects you, how well are you doing?'
Current Knee Pain | Baseline to Hours 2-6
  After completing a walk of approximately 50 feet, subjects will record their level of Current Knee Pain in the target knee on a 100-mm Visual Analog Scale (with anchors 0=no pain; 100=extreme pain) in response to the question, 'How do you estimate the amount of your study knee pain right now?'
WOMAC Stiffness Subscale | Baseline to Weeks 2, 4 and 6
  The WOMAC NRS3.1 OA Index is a validated, segregated, multidimensional, self-administered index with three independent dimensions: pain, physical function and stiffness. It is comprised of 24 questions to be answered by the subject. The pain subscale consists of 5 questions; the physical function subscale consists of 17 questions; and the joint stiffness subscale consists of 2 questions.
Pain on Movement (VAS, in-clinic) | Baseline to Weeks 2, 4 and 6
  Subjects will record their level of Pain on Movement in the target knee on a 100-mm VAS scale (with anchors 0=no pain; 100=extreme pain) in response to the question, 'How do you estimate the average amount of your study knee pain while moving during your daily activities within the last 24 hours?'
Pain on Movement (11-point NRS, diary) | Baseline through Week 6
  All evaluations will be on the 11-point Numerical Rating Scale (with anchors 0=no pain; 100=extreme pain) and in response to the following instructions: Please put an "X" over the one number below that best describes your average study knee pain while moving during your daily activities since you woke up this morning.
Use of Rescue Medication | Baseline through Week 6
  Subjects will record the amount, time/date and dose of Rescue Medication use throughout the trial.
Short Form 12v2 Health Survey | Baseline to Weeks 2, 4 and 6
  The SF-12v2 Health Survey is a multipurpose short-form (SF) general health survey comprised of 12 questions to measure functional health and well-being from the subject's perspective.

OTHER OUTCOMES:
Physical Examination: Number of subjects with clinically significant changes in Physical Examination in major body systems (HEENT, Neck, Cardiovascular, Abdominal, Respiratory, Musculoskeletal, Extremities Skin or Other) | Baseline through Week 8
Vital Signs: Change from Baseline in Heart Rate (beats per minute) | Baseline through Week 8
Vital Signs: Change from Baseline in Supine Diastolic Blood Pressure [mmHg] | Baseline through Week 8
Vital Signs: Change from Baseline in Supine Systolic Blood Pressure [mmHg] | Baseline through Week 8
Vital Signs: Change from Baseline in Body Temperature (axillary) [°C] | Baseline through Week 8
Vital Signs: Change from Baseline in respiration rate (respirations per minute) | Baseline through Week 8
Number of Adverse Events | Screening through Week 8
Number of Serious Adverse Events | Screening through Week 8
Number of Treatment Emergent Adverse Events | Baseline through Week 8
Percent of Subjects experiencing Adverse Events | Screening through Week 8
Percent of Subjects experiencing Serious Adverse Events | Screening through Week 8
Percent of Subjects experiencing Treatment Emergent Adverse Events | Baseline through Week 8
Safety Labs: Hematology | Baseline through Week 8
  Blood will be drawn for hematology laboratory analysis
Safety Labs: Chemistry | Baseline through Week 8
  Blood will be drawn for chemistry laboratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: William Cunningham, MD, FAAD, Study Chair — Cu-Tech, LLC
Locations (13):
- United States (13):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Avail Clinical Research, DeLand, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Sunrise Medical Research, Inc., Lauderdale Lakes, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - Miami Research Associates, LLC, South Miami, Florida
  - Best Clinical Trial, LLC, New Orleans, Louisiana
  - Healthcare Research Network, Inc., Hazelwood, Missouri
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Inc, Mt. Pleasant, South Carolina
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia